CLINICAL TRIAL: NCT00274651
Title: A Phase II Clinical Trial of PXD101 in Patients With Recurrent or Refractory Cutaneous and Peripheral T-Cell Lymphomas
Acronym: PXD101-CLN-6
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Enrollment stopped prior to reaching expected number of patients, study had accumulated sufficient data to allow a registration study in PTCL (PXD101-CLN-19)
Sponsor: Valerio Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PXD101-CLN-6
Record Dates: First submitted 2006-01-10; First posted 2006-01-11 (Estimated); Results first posted 2014-10-27 (Estimated); Last update posted 2015-07-28 (Estimated); Status verified 2015-07

CONDITIONS: Cutaneous T-Cell Lymphoma; Peripheral T-Cell Lymphoma; Non-Hodgkin's Lymphoma
Keywords: CTCL; PTCL; lymphoma; Non-Hodgkin's Lymphoma; Cutaneous T-Cell Lymphomas (CTCL); Peripheral T-Cell Lymphomas (PTCL); Other Types of Non-Hodgkin's Lymphoma; belinostat
MeSH Terms: conditions — Lymphoma, T-Cell, Cutaneous; Lymphoma, T-Cell, Peripheral; Lymphoma, Non-Hodgkin; Lymphoma | interventions — belinostat

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm A (Experimental): PXD101 1000 mg/m2 once daily for 5 days every 21 days
  Interventions: Drug: belinostat
- Arm B (Experimental): PXD101 1000 mg/m2 once daily for 5 days every 21 days
  Interventions: Drug: belinostat

INTERVENTIONS:
Drug: belinostat
  Other Names: PXD101

SUMMARY:
Open-label, non-randomized trial to assess the effectiveness of PXD101 in patients with recurrent or refractory cutaneous or peripheral and other types of T-cell lymphomas. PXD101 is a new, potent histone deacetylase (HDAC) inhibitor. Patients are treated with belinostat(PXD101) 1000 mg/m2 on days 1-5 of a 21 day cycle.

ELIGIBILITY:
Inclusion Criteria:

* Male or female with age > or = 18 years.
* Histologically confirmed diagnosis of cutaneous T-cell lymphoma (CTCL) or peripheral T-cell lymphoma (PTCL) or other T-cell non-Hodgkin's lymphoma (NHL).
* Must have failed at least one line of prior systemic therapy. No limitation in number of prior therapies. CTCL patients who are refractory or intolerant to oral Targretin are also eligible.
* The presence of measurable disease (defined as > or = 1 cm with radiographic imaging) for PTCL or stage 1B or greater disease for CTCL and assessable by the severity-weighted assessment tool (SWAT).
* Adequate bone marrow and hepatic function including the following:

  * Absolute neutrophil count > or = 1,000 cells/mm3, platelets > or = 40,000/mm3
  * Total bilirubin < or = 1.5 x upper normal limit or < or = 3 x upper normal limit if hepatic involvement
  * AST (SGOT) (aspartate aminotransferase), ALT (SGPT) (alanine aminotransferase) < or = 2.5 x upper normal limit (< or = 5 x upper normal limit if hepatic involvement)
  * Hemoglobin > or = 9.0 g/dL.
* Serum potassium within normal range.
* Karnofsky performance status > or = 70%.
* Estimated life expectancy > 3 months.
* Signed informed consent approved by the Institutional Review Board (IRB).

Exclusion Criteria:

* Anti-cancer therapies within 4 weeks of first PXD101 administration should be excluded unless toxicity from prior anti-cancer therapy has resolved or returned to baseline and cancer disease status warrants.
* Any use of investigational drugs within 4 weeks prior to study registration.
* Major surgery within 4 weeks of study drug administration.
* Prior allogeneic bone marrow transplant.
* A diagnosis of adult T-cell lymphoma/leukemia (ATLL) or precursor T-lymphoblastic lymphoma.
* Co-existing active infection or any co-existing medical condition likely to interfere with trial procedures. However, patients with progressing CTCL whose open skin lesions are frequently infected may not be excluded from this trial at the discretion of Investigators.
* Clinically significant cardiovascular disease including unstable angina pectoris, uncontrolled hypertension, and congestive heart failure related to primary cardiac disease, a condition requiring anti-arrhythmic therapy, history of sustained ventricular tachycardia, history of ventricular fibrillation or Torsade de Pointes, bradycardia (HR<50bpm) with or without a pacemaker, bifascicular block with a right bundle branch block and a left anterior block, ischemic or severe valvular heart disease, a myocardial infarction within 6 months or a left ventricular ejection fraction < 40% (by echocardiogram [ECHO] or multigated acquisition scan [MUGA]) within 3 months of study enrolment.
* A marked baseline prolongation of QT/QTc ((corrected) QT) interval, e.g., repeated demonstration of a QTc interval > 450 milliseconds (msec). Long QT Syndrome; the required use of concomitant medication on belinostat infusion days that may cause Torsade de Pointes.
* Renal insufficiency defined as a calculated creatinine clearance of < 45 mL/min/1.73 m2.
* A history of allergic reactions attributed to compounds of similar chemical or biological composition to PXD101 and L-arginine.
* Clinically significant central nervous system disorders with altered mental status or psychiatric disorders precluding understanding of the informed consent process and/or completion of the necessary studies.
* Patients requiring treatment for other malignant diseases or less than 5 years post-treatment completion for an invasive malignant disease (excluding non-melanotic skin cancers or cervical cancer in-situ). Patients with any history of melanoma should be excluded.
* Pregnant or breast-feeding women, and women of childbearing age and potential, who are not willing to use effective contraception. Male patients and/or their fertile female partners who are not willing to use contraceptives during the trial.
* Known infection with HIV, human T-cell leukemia virus type-1 (HTLV-1), hepatitis B or hepatitis C.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2006-01; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: e-mail contact via enquiries@topotarget.com, Study Director — Valerio Therapeutics
Locations (15):
- United States (8):
  - Leland Stanford Junior University, Stanford, California
  - Yale University School of Medicine, New Haven, Connecticut
  - Kansas City Cancer Center, Lenexa, Kansas
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Boston University Medical Center, Boston, Massachusetts
  - NYU Medical Center, New York, New York
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - MD Anderson Cancer Center, Houston, Texas
- France (2):
  - Hopitaux du Haut Leveque, Pessac
  - Hospital Purpan, Toulouse
- Universitatsklinikum Essen, Essen, Germany
- Israel (2):
  - Hadassah University Hospital Ein Kerem, Jerusalem
  - Rabin Medical Center, Petah Tikva
- Thailand (2):
  - Songklanagarind Hospital, Prince of Songkla University, Hat Yai
  - King Chulalongkorn Memorial Hospital, Patumwan

REFERENCES:
- [Derived] Foss F, Advani R, Duvic M, Hymes KB, Intragumtornchai T, Lekhakula A, Shpilberg O, Lerner A, Belt RJ, Jacobsen ED, Laurent G, Ben-Yehuda D, Beylot-Barry M, Hillen U, Knoblauch P, Bhat G, Chawla S, Allen LF, Pohlman B. A Phase II trial of Belinostat (PXD101) in patients with relapsed or refractory peripheral or cutaneous T-cell lymphoma. Br J Haematol. 2015 Mar;168(6):811-9. doi: 10.1111/bjh.13222. Epub 2014 Nov 17. PMID 25404094

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm A (CTCL, ITT Population); Arm B (PTCL, ITT Population): PXD101 1000 mg/m2 once daily for 5 days every 21 days
Period: Overall Study
Arm/Group | Arm A (CTCL, ITT Population) | Arm B (PTCL, ITT Population)
Started | 29 | 24
Completed | 1 | 4
Not Completed | 28 | 20
Not completed — Adverse Event | 6 | 3
Not completed — Lack of Efficacy | 13 | 6
Not completed — Death | 1 | 3
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Physician Decision | 8 | 7

BASELINE CHARACTERISTICS:
Population: Patients received PXD101, 1000 mg/m2/day over 30 minutes days 1-5 of a 21-day cycle. Patients with OR or stable disease were permitted to continue with PXD101 for up to 8 cycles or until progressive disease. Patients with PR or SD could continue therapy beyond 8 cycles until progression in consultation with Investigators and Sponsor.
Groups:
- CTCL (ITT Population): CTCL patients will receive 1000 mg/m2 of PXD101 IV
  belinostat: 1000 mg/m2 for 5 days every 21 days; IV
- PTCL (ITT Population): PTCL patients will receive 1000 mg/m2 of PXD101 IV
  belinostat: 1000 mg/m2 for 5 days every 21 days; IV
- Total: Total of all reporting groups
Arm/Group | CTCL (ITT Population) | PTCL (ITT Population) | Total
Number analyzed (Participants) | 29 | 24 | 53
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.1 (13.4) | 58.8 (15.9) | 61.7 (14.7)
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 12 | 12 | 24
  >=65 years | 17 | 12 | 29
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 7 | 22
  Male | 14 | 17 | 31
Region of Enrollment [Number; unit: participants]
  United States | 22 | 17 | 39
  France | 2 | 0 | 2
  Israel | 2 | 1 | 3
  Thailand | 2 | 6 | 8
  Germany | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate in Patients With Recurrent or Refractory Cutaneous T-cell Lymphoma (CTCL)
Description: Tumor response was assessed using Cheson (Cheson 2007) and SWAT criteria. The SWAT score represents the product of the percentage total body surface area (TBSA) involvement of each lesion type (patch, plaque, and tumor or ulceration), multiplied by a weighting factor.
Time Frame: throughout the study, or for a maximum of 2 years
Population: At termination OR was noted in 1/13 patients (Simon Stage 1). With 29 patients in the CTCL arm the demand for expansion to Simon Stage 2 lacked 5 patients and the study was stopped. Instead OR was done as secondary efficacy analysis (ITT and PP (per protocol)) with OR calculated without accounting for Simon design and with 95% confidence intervals
Groups:
- Arm A (CTCL, ITT Population): CTCL patients will receive 1000 mg/m2 of PXD101 IV
  belinostat: 1000 mg/m2 for 5 days every 21 days; IV
Arm/Group | Arm A (CTCL, ITT Population)
Number analyzed (Participants) | 0

2. Primary Outcome: Objective Response Rate in Patients With Recurrent or Refractory Peripheral T-cell Lymphoma (PTCL))
Description: Tumor response was assessed using the revised criteria of Cheson (Cheson 2007).Tumor assessments were done using conventional radiographic methods, e.g. CT or CT/PET.
Time Frame: throughout the study, or for a maximum of 2 years
Population: Primary efficacy analysis is based on the ITT analysis set, where the OR are calculated, and the proportion ± 80% CI (confidence interval) specified by Koyama & Chen (2008) are presented
Measure: Number; unit: percentage of patients with OR
Arm/Group | PTCL (ITT Population)
Number analyzed (Participants) | 24
percentage of patients with OR | 25

3. Secondary Outcome: Time to Progression
Description: Time to progression was defined as the interval between the first date of treatment and the first notation of disease progression.
Time Frame: throughout the study, or for a maximum of 2 years
Population: Time to Progression (ITT population) was estimated using the Kaplan-Meier method for CTCL and PTCL arms. As progression was not observed in six patients in Arm A and 10 patients in Arm B, a total of 37 patients progressed, and the the median time to progression and the full range (days) are presented.
Measure: Median (Full Range); unit: Days
Groups:
- Arm B (PTCL, ITT Population): PTCL patients will receive 1000 mg/m2 of PXD101 IV
  belinostat: 1000 mg/m2 for 5 days every 21 days; IV
Arm/Group | Arm A (CTCL, ITT Population) | Arm B (PTCL, ITT Population)
Number analyzed (Participants) | 23 | 14
Days | 43 [15 to 304] | 82 [9 to 890]

4. Secondary Outcome: Time to Response
Description: Time to response was defined as the interval between the first date of treatment and the first notation of response.
Time Frame: throughout the study, or for a maximum of 2 years
Population: Time to response (ITT population) was estimated using the Kaplan-Meier method for CTCL and PTCL arms. For 4 patients with CTCL and 6 patients with PTCL, response was recorded. The median time to response and the full range (days) are presented.
Measure: Median (Full Range); unit: Days
Arm/Group | Arm A (CTCL, ITT Population) | Arm B (PTCL, ITT Population)
Number analyzed (Participants) | 4 | 6
Days | 40 [15 to 176] | 100 [9 to 431]

5. Secondary Outcome: Duration of Response
Description: Duration of response was defined as the time from first notation of response until the time of first notation of disease progression.
Time Frame: throughout the study, or for a maximum of 2 years
Population: Duration of response (ITT population) was estimated by Kaplan-Meier method for CTCL/PTCL arms. 2 CTCL and 2 PTCL patients did not progress and were censored. Median duration of response and full range (days) are presented for 2 patients with CTCL and 4 patients with PTCL. The 2 CTCL patients being evaluable had response durations of 56 and 129 days
Measure: Median (Full Range); unit: Days
Arm/Group | Arm A (CTCL, ITT Population) | Arm B (PTCL, ITT Population)
Number analyzed (Participants) | 2 | 4
Days | 83 [56 to 129] | 109 [7 to 460]

6. Post Hoc Outcome: Objective Response Rate in Patients With Recurrent or Refractory Cutaneous T-cell Lymphoma (CTCL)
Description: as for outcome 1
Time Frame: throughout the study, or for a maximum of 2 years
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Arm A (CTCL, ITT Population)
Number analyzed (Participants) | 29
participants | 4

ADVERSE EVENTS:
Time Frame: Throughout study, up to 4 weeks after last drug administration
Description: Follow-up of the AE (adverse event) was required during the study and after completion, withdrawal or discontinuation of the study if the event was still ongoing. The Investigator was to continuously monitor patients with AEs until the event had returned to baseline or ≤ Grade 1 or until the patient started another type of antineoplastic therapy.
Arm/Group | Arm A (CTCL, ITT Population) | Arm B (PTCL, ITT Population)
Serious Adverse Events (participants affected / at risk) | 7/29 | 8/24
Other Adverse Events (participants affected / at risk) | 29/29 | 23/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A (CTCL, ITT Population) (N=29) | Arm B (PTCL, ITT Population) (N=24)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Disease progression (General disorders) | 1 (1) | 1 (1)
Staphylococcal skin infection (Infections and infestations) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 1 (3)
Gait disturbance (General disorders) | 1 (1) | 0 (0)
Oedema peripheral (General disorders) | 1 (1) | 0 (0)
Apraxia (Nervous system disorders) | 1 (1) | 0 (0)
Jugular vein thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Implant site abscess (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 2 (2) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Ventricular fibrillation (Cardiac disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Ileus paralytic (Gastrointestinal disorders) | 0 (0) | 1 (1)
Catheter related infection (Infections and infestations) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A (CTCL, ITT Population) (N=29) | Arm B (PTCL, ITT Population) (N=24)
Fatigue (General disorders) | 6 (11) | 8 (11)
Pyrexia (General disorders) | 5 (9) | 6 (16)
Infusion site pain (General disorders) | 6 (6) | 3 (3)
Oedema peripheral (General disorders) | 6 (7) | 1 (1)
Injection site reaction (General disorders) | 0 (0) | 5 (9)
Asthenia (General disorders) | 1 (1) | 2 (2)
Chest pain (General disorders) | 3 (3) | 0 (0)
Chills (General disorders) | 3 (3) | 0 (0)
Disease progression (General disorders) | 1 (1) | 2 (2)
Gait disturbance (General disorders) | 3 (3) | 0 (0)
Oedema (General disorders) | 1 (1) | 2 (2)
Nausea (Gastrointestinal disorders) | 17 (29) | 16 (32)
Constipation (Gastrointestinal disorders) | 5 (5) | 9 (10)
Vomiting (Gastrointestinal disorders) | 8 (14) | 6 (19)
Diarrhoea (Gastrointestinal disorders) | 4 (4) | 5 (10)
Dyspepsia (Gastrointestinal disorders) | 3 (3) | 3 (4)
Abdominal pain (Gastrointestinal disorders) | 3 (3) | 2 (4)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 3 (4)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 2 (2)
Dizziness (Nervous system disorders) | 6 (7) | 5 (8)
Headache (Nervous system disorders) | 6 (6) | 1 (1)
Dysgeusia (Nervous system disorders) | 3 (3) | 1 (1)
Hypoparaesthesia (Nervous system disorders) | 3 (3) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 3 (3) | 5 (5)
Hypokalaemia (Metabolism and nutrition disorders) | 3 (5) | 4 (9)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 4 (4)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
Pruritus (Skin and subcutaneous tissue disorders) | 7 (8) | 2 (2)
Rash (Skin and subcutaneous tissue disorders) | 4 (5) | 3 (3)
Skin exfoliation (Skin and subcutaneous tissue disorders) | 4 (4) | 0 (0)
Alanine aminotransferase increased (Investigations) | 2 (2) | 2 (3)
Aspartate aminotransferase increased (Investigations) | 2 (2) | 2 (2)
Blood alkaline phosphatase increased (Investigations) | 1 (1) | 3 (3)
Blood lactate dehydrogenase increased (Investigations) | 3 (3) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 3 (3) | 2 (2)
Cellulitis (Infections and infestations) | 2 (2) | 2 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 5 (6) | 5 (5)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (3) | 3 (4)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 2 (3)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (2)
Flushing (Vascular disorders) | 1 (1) | 4 (4)
Phlebitis (Vascular disorders) | 3 (3) | 1 (1)
Tachycardia (Cardiac disorders) | 1 (2) | 3 (6)
Eosinophilia (Blood and lymphatic system disorders) | 2 (3) | 1 (1)
Lymphadenopathy (Blood and lymphatic system disorders) | 2 (3) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 3 (4)
Confusional state (Psychiatric disorders) | 2 (2) | 2 (2)
Insomnia (Psychiatric disorders) | 1 (1) | 2 (4)
Mucosal inflammation (General disorders) | 2 (2) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 2 (3)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 2 (2)
Hypomagnesaemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Blood creatinine increased (Investigations) | 2 (3) | 0 (0)
Blood magnesium decreased (Investigations) | 0 (0) | 2 (2)
Blood uric acid increased (Investigations) | 2 (2) | 0 (0)
Body temperature increased (Investigations) | 2 (2) | 0 (0)
Herpes simplex (Infections and infestations) | 2 (2) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 2 (2)
Sepsis (Infections and infestations) | 2 (2) | 0 (0)
Skin infection (Infections and infestations) | 2 (2) | 0 (0)
Tinea pedis (Infections and infestations) | 2 (2) | 0 (0)
Muscle spams (Musculoskeletal and connective tissue disorders) | 2 (3) | 1 (2)
Neck pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Hypotension (Vascular disorders) | 2 (2) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
Vertigo (Ear and labyrinth disorders) | 2 (3) | 0 (0)
Hypersensitivity (Immune system disorders) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less